CLINICAL TRIAL: NCT06382077
Title: Determination of the Frequency and Affecting Factors of Chronic Postsurgical Pain After Cardiac Surgery: A Multicenter, Observational Study
Brief Title: Chronic Post Surgical Pain-Cardiac
Acronym: CPSP-Cardiac
Status: Active, not recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Coordinating Investigator, Ondokuz Mayıs University
Other Study IDs: CPSP5502
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Post-surgical Pain
Keywords: cardiac anesthesia; chronic post-surgical pain; nerve blocks
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CPSP-Cardiac is a large, multi-center, observational study with the aim to investigate the incidence of chronic pain in the 3rd month postoperatively in cardiac surgery and its affecting factors.

DETAILED DESCRIPTION:
Cardiovascular diseases pose a significant global health concern, particularly among the elderly population, leading to a surge in surgical interventions. Enhanced Recovery After Surgery (ERAS®) protocols, specifically ERAS® Cardiac, target improved perioperative pain management to optimize patient outcomes. Effective pain control aims to alleviate acute discomfort, prevent chronic pain development, facilitate early mobilization, reduce hospital stays, and enhance patient satisfaction and functional recovery. While pain intensity peaks within the initial days following cardiac surgery and gradually subsides, inadequate acute pain management can predispose patients to chronic pain, impairing their quality of life. Multimodal opioid-sparing analgesia strategies are recommended, with recent advancements in ultrasound-guided regional anesthesia techniques showing promise in enhancing acute pain relief and reducing opioid consumption, particularly through truncal fascial plane blocks and parasternal blocks. However, the impact of these techniques on chronic postsurgical pain remains incompletely understood. This multicenter study aims to investigate the incidence of chronic postsurgical pain following cardiac surgery, exploring the influence of various factors and their implications on patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients will be undergoing a first-time cardiac surgery involving a median sternotomy, including coronary artery bypass grafting (CABG) and all open-heart procedures, such as valvular repairs/replacement.
* patients between the ages of 18-80 years
* American Society of Anesthesiologists (ASA) Physical Status score of II-III
* patients will also sign the written informed consent form

Exclusion Criteria:

* patients scheduled for minimally invasive cardiac surgery,
* patients with BMI>40,
* patients who undergone thoracotomy,
* patients with alcohol and drug addiction,
* patients with severe dysfunction in a significant organ (e.g., presence of severe hepatic and renal disease),
* patients who undergone emergency and redo surgeries,
* patients who cannot be extubated within the first 8 hours postoperatively,
* patients have a severe psychiatric diseases such as psychosis or dementia that restrict cooperation with the patient (patients who cannot evaluate verbal numerical pain scales),
* patients who are pregnant and breastfeeding,
* patients who cannot be reached by phone during the postoperative follow-up periods
* patients who cannot communicate in the native language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of 1176 cardiac surgery patients will be recruited from participating hospital sites. Patients eligible for our study will be undergoing a first-time cardiac surgery involving a median sternotomy, including CABG and all open-heart procedures, such as valvular repairs/replacement
Sampling Method: Probability Sample
Enrollment: 2442 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic postsurgical pain | Postoperative 3rd and 6th months
  The incidence of chronic postsurgical pain (CPSP) in the third month following cardiac surgery along with identifying the factors that influence it. CPSP as pain that (A) emerges after surgery, (B) is distinct from pre-procedural pain, (C) is not caused by other factors, and (D) persists for at least three months.

SECONDARY OUTCOMES:
Postoperative opioid consumption in the first 24 hours | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured.
Postoperative pain scores | Postoperative day 1
  Pain at rest and during activity (coughing and deep breathing) will be assessed by numerical rating scale (NRS) scores at 0, 3, 6, 12, and 24 hours after extubation. The NRS is an 11-point numeric scale that ranges from 0 to 10. The NRS is an 11-point scale consisting of integers from 0 to 10: 0 indicates "no pain" and 10 indicates "the worst pain ever possible."
The incidences of postoperative nausea and vomiting | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, and 24 hours after extubation. The PONV scale is 0 = none, 1 = mild nausea, 2 = moderate nausea, 3 = vomiting once, and 4 = vomiting more than once
The number of patients with side effects and complications | The time from surgery to the time of discharge to the home; an average of 14 days
  The number of patients have any side effects and complications will be recorded.
Time to extubation | Postoperative Day 1
  After the operation, the time until the patient is extubated will be recorded.
Length of stay in the intensive care unit | The time from admission to the ICU to the time of discharge to the hospital ward; during the hospital stay, an average of 7 days
  Total duration of stay in intensive care unit (ICU) will be recorded
Length of stay in the hospital | Measured in days admitted in the hospital, an average of 14 days
  Their stay in the hospital will be recorded.
Chronic pain status at 3 and 6 months | 90 and 180 days after surgery
  After discharge, patients will be contacted at 3 and 6 months. Pain intensity and status will be assessed using the Brief Pain Inventory-Short Form, and the character of pain will be evaluated using the Leeds Assessment of Neuropathic Signs and Symptoms Pain Questionnaire score.
Psychological assessment | 90 and 180 days after surgery
  The patient's anxiety and depression status will be assessed using the Hospital Anxiety and Depression Scale.
Quality of life assessment | 90 and 180 days after surgery
  Pain Self-Efficacy Questionnaire will be used to assess the influence of chronic pain on the individual's daily life.
Postoperative complications at 3 and 6 months | 90 and 180 days after surgery
  The severity of complications will be evaluated using the 'Clavien-Dindo' classification. Additionally, the 'Comprehensive Complication Index' (https://www.cci-calculator.com/cciCalculator) will be used to evaluate the patient's overall postoperative morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan DOST, Assoc.Prof, Study Director — Ondokuz Mayıs University
Locations (29):
- Turkey (Türkiye) (29):
  - Ondokuz Mayis University, Samsun, Atakum
  - Adiyaman Üniversitesi, Adıyaman
  - Ankara University, Ankara
  - Bilkent City Hospital, Ankara
  - Hacettepe Üniversitesi, Ankara
  - Akdeniz University, Antalya
  - Antalya Eah, Antalya
  - Bursa City Hospital, Bursa
  - Bursa Yuksek Ihtisas Eah, Bursa
  - Uludağ Üniversitesi, Bursa
  - Canakkale University, Çanakkale
  - Hitit University, Çorum
  - Denizli Dh, Denizli
  - Ataturk University, Erzurum
  - Süleyman Demirel Üniversitesi, Isparta
  - Acibadem Atasehir Hospital, Istanbul
  - Basahsehir Cam and Sakura Hospital, Istanbul
  - Istanbul University, Istanbul
  - Kartal Kosuyolu Eah, Istanbul
  - Marmara University, Istanbul
  - Medipol Mega Hospital, Istanbul
  - İzmir Katip Çelebi University, Izmir
  - Kocaeli University, Kocaeli
  - Kocaeli Şehir Hastanesi, Kocaeli
  - Mersin University, Mersin
  - Muğla Eah, Muğla
  - Samsun University, Samsun
  - Karadeniz Teknik University, Trabzon
  - Trabzon Ahi Avran Eah, Trabzon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maessen T, Korir N, Van de Velde M, Kennes J, Pogatzki-Zahn E, Joshi GP; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy. Pain management after cardiac surgery via median sternotomy: A systematic review with procedure-specific postoperative pain management (PROSPECT) recommendations. Eur J Anaesthesiol. 2023 Oct 1;40(10):758-768. doi: 10.1097/EJA.0000000000001881. Epub 2023 Jul 19. PMID 37501517
- [Background] Xiao MZX, Khan JS, Dana E, Rao V, Djaiani G, Richebe P, Katz J, Wong D, Clarke H. Prevalence and Risk Factors for Chronic Postsurgical Pain after Cardiac Surgery: A Single-center Prospective Cohort Study. Anesthesiology. 2023 Sep 1;139(3):309-320. doi: 10.1097/ALN.0000000000004621. PMID 37192204
- [Background] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838